CLINICAL TRIAL: NCT05906901
Title: Effects of Osteopathic Treatment in Patients With Tension Type Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OST1-009
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The investigator will perform a cranial listening technique.
  Interventions: Other: Cranial listening technique
- Suboccipital muscles inhibition (Experimental): The investigator will perform a suboccipital muscles inhibition technique.
  Interventions: Other: Suboccipital muscles inhibition technique

INTERVENTIONS:
Other: Cranial listening technique — 5 minutes
  Arms: Control Group
Other: Suboccipital muscles inhibition technique — 6 minutes
  Arms: Suboccipital muscles inhibition

SUMMARY:
The aim of this study is to evaluate the effects of the suboccipital muscles inhibition technique on patients suffering from tension-type headaches.

DETAILED DESCRIPTION:
The tension-type headache is a recurrent condition with a high financial repercussion in Portugal. Their side effects often impact daily activities, reducing the quality of life of the patients.

In several studies, the excessive tension of the suboccipital muscles are usually referred as a cause of tension-type headache, since they can exert tension on the dura mater through the myodural bridge.

ELIGIBILITY:
Inclusion Criteria:

They must have tension-type headache, that is, a headache with:

* a duration of at least 30 min to days, with or without an break;
* must have at least two of the following four characteristics:

  1. bilateral location
  2. pressure or squeezing quality (non throbbing)
  3. weak or moderate intensity
  4. not aggravated by routine physical activity such as walking or climbing stairs;
* must have both of the following criteria:

  1. only one of the following: photophobia, phonophobia, or mild nausea
  2. absence of moderate or severe nausea or vomiting.

Exclusion Criteria:

* They can't be on antibiotics, antivirals, or antidepressants;
* They can't have neurological problems;
* They shouldn't have any absolute contraindication for the osteopathic maneuvers;
* They can't have acute pathologies (ex: infection) or serious (ex: cancer);
* They can't have fractures in the skull, cervical spine or high dorsal spine (up to D4);
* They can't be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency | One month after first intervention
  Measured by monthly counting.
Intensity | One month after first intervention
  Measured by visual analogue scale (VAS). It goes from 0 to 10, 0 being the minimum pain intensity and 10 the maximum pain intensity.
Impact on quality of life questionnaire | one month after first intervention
  Measured by questionnaire. The questionnaire attribuates a score after answering six questions. The lowest score a participant can obtain is 36, which corresponds to the lowest impact on quality of life. The highest score a participant can obtain is 78, which corresponds to the highest impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Natália, Principal Investigator — Escola Superior da Saúde do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276